CLINICAL TRIAL: NCT02615431
Title: the Influence of MitraClip on Apnoea Asleep
Acronym: MiClAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-060
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2015-11

CONDITIONS: Sleep Apnoea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MitraClip Intervention: the influence of MitraClip on Apnoea Asleep
  Interventions: Other: MitraClip Intervention

INTERVENTIONS:
Other: MitraClip Intervention

SUMMARY:
The aim of the present study is to influence the central and obstructive sleep apnoea in patients with severe mitral insufficiency by an interventional MitraClip examination to evaluate.

ELIGIBILITY:
Inclusion Criteria:

* patient suffer on severe symptomatical mitral insufficience
* male and female patients is planned an interventional MitraClip examination
* Dyspnea with a NYHA (New York Heart Association) II - III
* an high logistic Euro-Score (> 20)
* no execution of surgical intervention because of relevant comorbidities

Exclusion Criteria:

* younger than 18 years
* pregnancy and breast-feeding
* persons without mental ability of capacity to understand and follow the instructions of the investigator
* persons in dependence from the sponsor or working with the sponsor
* participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female patients is planned an interventional MitraClip examination
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Apnoea-Hypopnoea-Index | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, MD, Principal Investigator — Uniklinik RWTH Aachen, Med. Klinik I
Locations (1):
- University Hospital RWTH Aachen, Department of Medical Clinic I, Aachen, Germany